CLINICAL TRIAL: NCT01258361
Title: Echocardiographic Assessment of Volume Variation Secondary to Preoperative Fasting
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2010/LM-03; 2010-A01275-34 (Other: ANSM)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Hypovolemia
Keywords: preoperative fasting
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: Patients will be recruited during anesthesia consultations carried out before programmed pelvic or visceral surgeries.
  Interventions: Procedure: echocardiography

INTERVENTIONS:
Procedure: echocardiography — Echocardiography is performed for all patients

SUMMARY:
The primary objective of this study is to demonstrate that preoperative fasting does not increase the rate of lowered blood volume (defined by a variation of 15% ΔITV during a leg lift) in patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is ASA (American Society of Anesthesiologists) class I, II or III
* The patient has not been fasting for more than 6 hours at the time of inclusion
* The patient is schelduled for a gynecological or visceral surgery

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding
* The patient is ASA class IV
* The patient has insulin dependent diabetes
* The patient has a cardiac or respiratory dysfunction
* The patient has a heart rhythm disorder
* The patient has renal insufficiency with dialysis
* The patient is being treated with diuretics
* The patient has had a bowel preparation
* Emergency surgery
* Outpatient surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited during anesthesia consultations carried out before programmed gynecological or visceral surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04-13 (Actual); Study Completion 2011-04-13 (Actual)

PRIMARY OUTCOMES:
The presence / absence of a hypovolemia following preoperative fasting | 1 day
  Hypovolemia is determined by the % change in the subaortic velocity time integral during a leg lift before and after fasting: a 15% decrease is considered as a "presence".

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Muller, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France

REFERENCES:
- [Result] Muller L, Briere M, Bastide S, Roger C, Zoric L, Seni G, de La Coussaye JE, Ripart J, Lefrant JY. Preoperative fasting does not affect haemodynamic status: a prospective, non-inferiority, echocardiography study. Br J Anaesth. 2014 May;112(5):835-41. doi: 10.1093/bja/aet478. Epub 2014 Feb 3. PMID 24496782